CLINICAL TRIAL: NCT03565367
Title: A Pilot Study to Assess Lactate and Bicarbonate Detection Within Malignant Brain Tumors Using [1-13C]-Pyruvate DNP Magnetic Resonance Spectroscopy (MRS)
Brief Title: Hyperpolarized Carbon C 13 Pyruvate Magnetic Resonance Spectroscopic Imaging in Detecting Lactate and Bicarbonate in Participants With Central Nervous System Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daniel M. Spielman (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Daniel M. Spielman, Professor of Radiology, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-39845; NCI-2018-01122 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB-39845 (Other: Stanford IRB); BRN0036 (Other: OnCore); R01CA245097-01A1 (NIH)
Record Dates: First submitted 2018-06-11; First posted 2018-06-21 (Actual); Results first posted 2023-12-18 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-11

CONDITIONS: Malignant Central Nervous System Neoplasm; Metastatic Malignant Neoplasm in the Central Nervous System
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Gadolinium; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Volunteers (Experimental): Participants undergo MRI over 45 minutes at baseline. Participants then receive hyperpolarized carbon C 13 pyruvate IV over 30-40 seconds. Within 1 minute, participants undergo MRSI over 3 minutes and MRI over 10 minutes.
  Interventions: Drug: Hyperpolarized Carbon C 13 Pyruvate; Procedure: Magnetic Resonance Imaging; Procedure: Magnetic Resonance Spectroscopic Imaging
- Known CNS Malignancy (Experimental): Participants undergo MRI over 45 minutes at baseline. Participants then receive hyperpolarized carbon C 13 pyruvate IV over 30-40 seconds. Within 1 minute, participants undergo MRSI over 3 minutes and MRI over 10 minutes (participants may receive gadolinium at the discretion of the protocol director).
  Interventions: Other: Gadolinium; Drug: Hyperpolarized Carbon C 13 Pyruvate; Procedure: Magnetic Resonance Imaging; Procedure: Magnetic Resonance Spectroscopic Imaging

INTERVENTIONS:
Other: Gadolinium — gadolinium enhanced MRI
  Other Names: Gd
  Arms: Known CNS Malignancy
Drug: Hyperpolarized Carbon C 13 Pyruvate — Given IV
  Other Names: Hyperpolarized 13C-Pyruvate; Hyperpolarized Pyruvate (13C)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Magnetic Resonance Spectroscopic Imaging — Undergo MRSI
  Other Names: 1H- Nuclear Magnetic Resonance Spectroscopic Imaging; 1H-nuclear magnetic resonance spectroscopic imaging; Magnetic Resonance Spectroscopy; MRS; MRS Imaging; MRSI; Proton Magnetic Resonance Spectroscopic Imaging

SUMMARY:
This early phase I trial studies how well hyperpolarized carbon C 13 pyruvate magnetic resonance imaging works in detecting lactate and bicarbonate in participants with central nervous system tumors. Hyperpolarized carbon C 13 pyruvate magnetic resonance imaging may be used to measure the metabolic state of malignant brain tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety of intravenous (IV) injection of hyperpolarized carbon C 13 pyruvate (hyperpolarized [1-13C] pyruvate) for magnetic resonance imaging (MRI).

II. To assess the frequency and sensitivity with which lactate and bicarbonate signals can be detected in malignant brain tumors after IV injection of hyperpolarized [1-13C] pyruvate.

OUTLINE:

Participants undergo MRI over 45 minutes at baseline. Participants then receive hyperpolarized carbon C 13 pyruvate IV over 30-40 seconds. Within 1 minute, participants undergo magnetic resonance spectroscopic imaging (MRSI) over 3 minutes and MRI over 10 minutes (participants may receive gadolinium at the discretion of the protocol director).

After completion of study, participants are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a known diagnosis of central nervous system (CNS) malignancy, including metastases, with known enhancement on magnetic resonance (MR) who are otherwise eligible to undergo MRI
* Glomerular filtration rate (GFR) > 30 ml/min
* No allergy to gadolinium
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Refusal to have an IV placed for injection
* Acute major illness (e.g., unstable angina, etc.) or other condition that makes participation unsafe, per the investigator?s judgement
* Total bilirubin > 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 2.5 x ULN
* Gamma-glutamyltransferase (GGT) > 2.5 x ULN
* Pregnant or breast-feeding
* Cardiovascular risk, including:

  * Poorly controlled hypertension, defined as either systolic > 170 or diastolic > 110
  * Congestive heart failure
  * Myocardial infarction within the past year
  * QT prolongation, defined as pretreatment corrected QT interval (QTc) > 440 msec in males or > 460 msec in females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Recht, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Volunteers: Participants undergo MRI over 45 minutes at baseline, then receive hyperpolarized carbon C 13 pyruvate IV over 30-40 seconds. Within 1 minute, participants undergo MRSI over 3 minutes and MRI over 10 minutes.
- Known CNS Malignancy: Participants undergo MRI over 45 minutes at baseline, then receive hyperpolarized carbon C 13 pyruvate IV over 30-40 seconds. Within 1 minute, participants undergo MRSI over 3 minutes and MRI over 10 minutes (participants may receive gadolinium at the discretion of the protocol director).
Period: Overall Study
Arm/Group | Healthy Volunteers | Known CNS Malignancy
Started | 7 | 2
Received Interventions | 3 | 2
Completed | 3 | 2
Not Completed | 4 | 0
Not completed — No scan due to technical issues | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteers | Known CNS Malignancy | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 2 or Higher Toxicities
Description: The measurement of this drug is the number of participants with Grade 2 or higher related adverse events (except for asymptomatic lab increases)
Time Frame: 2 days (+/-2) after the scan
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers | Known CNS Malignancy
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

2. Other Pre Specified Outcome: Lactate and Bicarbonate Production in Tumor and Normal Brain Tissue
Description: The outcome is defined as the number of participants with hyperpolarized carbon C 13 pyruvate magnetic resonance signal detection above background noise level of both lactate and bicarbonate in all tumors screened.
Time Frame: Imaging timepoint (up to 15 minutes to obtain scan)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 4 days
Arm/Group | Healthy Volunteers | Known CNS Malignancy
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 2/3 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Volunteers (N=3) | Known CNS Malignancy (N=2)
Anosmia (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/67/NCT03565367/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/67/NCT03565367/ICF_002.pdf